CLINICAL TRIAL: NCT03342326
Title: Lexical Priming by Music in Alzheimer's Disease and Healthy Aging
Acronym: PriMus
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: failure to recruit
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1708117; 2017-A02686-47 (Other: ANSM)
Record Dates: First submitted 2017-11-10; First posted 2017-11-14 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Alzheimer Disease
Keywords: Lexical priming; Healthy Aging
MeSH Terms: conditions — Alzheimer Disease | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patient with Alzheimer's Disease (Other): 1. Exposure to familiar songs : a) Words and Music (sing condition), b) Words only (spoken condition) and c) Music only (instrumental condition) After each song : rate the popularity of the song on a scale of 1 to 5.
  2. Music Experience Questionnaire : questions about the past music training
  3. Implicit tasks memory : a) Completion of trigrams : freely complete the first 3 letters of a word. b) lexical decision : judge whether an audibly presented sound sequence is a word existing in the French language or not.
  Interventions: Other: Exposure to familiar songs; Other: Music Experience Questionnaire; Other: Implicit tasks memory
- healthy volunteer (Other): 1. Exposure to familiar songs : a) Words and Music (sing condition), b) Words only (spoken condition) and c) Music only (instrumental condition) After each song : rate the popularity of the song on a scale of 1 to 5.
  2. Music Experience Questionnaire : questions about the past music training
  3. Implicit tasks memory : a) Completion of trigrams : freely complete the first 3 letters of a word. b) lexical decision : judge whether an audibly presented sound sequence is a word existing in the French language or not.
  4. For volunteer over 65 years : Mini Mental State Examination, 5 words by Dubois and fluence verbal test
  Interventions: Other: Exposure to familiar songs; Other: Music Experience Questionnaire; Other: Implicit tasks memory; Other: Questionnaires

INTERVENTIONS:
Other: Exposure to familiar songs — 3 conditions : a) Words and Music (sing condition), b) Words only (spoken condition) and c) Music only (instrumental condition) After each song : rate the popularity of the song on a scale of 1 to 5.
Other: Music Experience Questionnaire — questions about the past music training
Other: Implicit tasks memory — 2 tests : a) Completion of trigrams : freely complete the first 3 letters of a word.
  b) lexical decision : judge whether an audibly presented sound sequence is a word existing in the French language or not.
Other: Questionnaires — Mini Mental State Examination, 5 words by Dubois and fluence verbal test
  Arms: healthy volunteer

SUMMARY:
While verbal memory is quickly reached in the wake of Alzheimer's disease, the musical memory remains preserved until a late stage of the disease. This observation encouraged the development of music-based therapies in the management of neurocognitive and behavioral disorders that characterize Alzheimer's disease. In order to develop rehabilitation programs that effectively target cognitive functions to stimulate, it is necessary to understand the mechanisms underlying this beneficial effect of music on cognition.

DETAILED DESCRIPTION:
The investigators study the stimulation by the song, material integrating language and music, and having an autobiographical value. The investigators measure the lexical priming capacity of the song, that is, its ability to activate and maintain lexical and semantic representations, which are threatened with alteration in the course of the disease.

This lexical priming effect by song is measured in patients with mild Alzheimer's disease and healthy volunteers during a single test session. In the first phase of the session, participants are exposed to familiar songs, presented in sung, spoken or instrumental form, whose popularity they evaluate. In the second phase, they perform two implicit memory tasks: a trigram completion task and a lexical decision task. These tests measure the facilitation of the processing of words evoked by songs in relation to words unrelated to songs, reflecting a "long-term" memory update of mnemic traces of primed words.

ELIGIBILITY:
Inclusion Criteria for patients :

* Presence of diagnostic criteria for Alzheimer's disease
* Age ≥ 65 years
* MMSE (Mini-mental state Examination) ≥ 20

Exclusion Criteria for patient :

* Unstable clinical presentation or language presentation in the foreground
* Cognitive disorder of etiology different from that of Alzheimer's disease

Inclusion Criteria for volunteers :

* Age ≥ 18 years
* Absence of neurological or psychiatric antecedents
* For those aged 65 or over: MMSE (Mini-mental state Examination) greater than or equal to 27; non-pathological performance against the 5 words of Dubois and the verbal fluency test.

Exclusion Criteria for volunteers :

* Visual or auditory disorders insufficiently corrected
* Oral or written expression in French insufficient to carry out tests
* Consumption of psychotropic drugs not stabilized

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2019-05-29 (Actual); Study Completion 2019-05-29 (Actual)

PRIMARY OUTCOMES:
Reaction time difference for the treatment of words that have been presented in sing condition in the exposure phase versus words presented in spoken condition. | Day 1

SECONDARY OUTCOMES:
Reaction time difference for processing words associated with songs presented by their melody alone versus new words (not presented in the exhibition phase). | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No